CLINICAL TRIAL: NCT05605106
Title: Addiction and Correlation With in Hospital Outcomes of Patients Presenting With Acute Coronary Syndrome Regarding to TIMI Flow and LV Function
Brief Title: Addiction and Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Amir Zaky Habib, resident doctor, Assiut University
Other Study IDs: addict ACS pts
Record Dates: First submitted 2022-10-28; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Acute Coronary Syndrome; Addiction
MeSH Terms: conditions — Acute Coronary Syndrome; Behavior, Addictive | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- addict patients presenting with acute coronary syndrome
  Interventions: Diagnostic Test: speckle tracking echocardiography; Procedure: Percutaneous coronary intervention
- non addict patients presenting with acute coronary syndrome
  Interventions: Diagnostic Test: speckle tracking echocardiography; Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Diagnostic Test: speckle tracking echocardiography — Speckle tracking is a recent development in image processing that uses proprietary software to automatically determine the movements of these points, which appear sonographically as "speckles," within the myocardium over time. Tracking the movements of these speckles throughout the cardiac cycle yields positive values when the two points are moving away from one another, as in diastole, and negative values when they are moving towards one another, as in systole
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention refers to a family of minimally invasive procedures used to open clogged coronary arteries (those that deliver blood to the heart). By restoring blood flow, the treatment can improve symptoms of blocked arteries, such as chest pain or shortness of breath.

SUMMARY:
the study aims to

1. identify the effect of addiction on TIMI flow in patients presented with acute coronary syndrome.
2. identify the effect of addiction on outcomes of medical treatment of patients presenting with acute coronary syndrome.
3. identify the relation between addiction and LV function.
4. detect the effect of duration of addiction on myocardial infarction lesion and outcomes of pci.

DETAILED DESCRIPTION:
substance abuse has been increasing nationally, yet its potential cardiovascular consequences are not fully understood.

There are limited data on the true prevalence of substance abuse in individuals who experience a myocardial infarction .

myocardial infarction is one of the most common diseases with high mortality and morbidity in human beings. There are many known risk factors in Coronary Artery Disease like; old age, male gender, cigarette smoking, hypertension, diabetes mellitus and hyperlipidemia .

Though, few studies have investigated the effect of addiction on coronary artery disease. Some studies reported harmful effects of addiction including opioid ,cocaine ,amphetamine and marijuana on the cardiovascular system . Some other studies did not find any association between drug addiction and coronary artery disease .

Thrombolysis in Myocardial Infarction (TIMI) coronary grade flow is an established, validated score to assess the epicardial perfusion on coronary angiography. TIMI flow grade 0 represents total occlusion, while TIMI flow grade 3 represents normal epicardial perfusion . Previous studies have demonstrated that patients with low grade TIMI flow prior to percutaneous coronary intervention (PCI) have a less favorable outcome. Preprocedural TIMI flow has been found to be an independent predictor of survival in patients with acute myocardial infarction , and has also been shown to predict final infarct size .

In the past decade, a new echocardiographic technique known as strain has been used to make more accurate assessments of the contractile state of the heart. Strain echocardiography has been used in a wide range of cardiovascular conditions including HF and acute coronary syndromes .Unlike conventional techniques of determining systolic function that rely on visual assessment of wall motion and changes in volume, strain echocardiography measures actual tissue deformation within the myocardium. Conceptually, strain can be thought of as a way to determine the movement between two points as if those two points are connected by a string. The physical definition of strain is the relative change in length of a material related to its original length.

Speckle tracking is a recent development in image processing that uses proprietary software to automatically determine the movements of these points, which appear sonographically as "speckles," within the myocardium over time. Tracking the movements of these speckles throughout the cardiac cycle yields positive values when the two points are moving away from one another, as in diastole, and negative values when they are moving towards one another, as in systole. Speckle tracking obviates the need for Doppler-based imaging technologies to calculate strain, which have proved to be challenging due to their angle-dependency .

LV strain on 2D echocardiography has been well studied in patients with ACS. For patients with ST-segment elevation MI , LV strain has been shown to be an important predictor of post-discharge adverse outcomes. .LV strain can also help discriminate which patients will successfully recover LV function and which patients will develop adverse LV remodeling .Moreover, decreased LV strain within 24 hours of revascularization for acute MI can reliably predict which patients are more likely to achieve a composite end-point of any of the following: all-cause mortality, hospitalization with re-infarction, HF, or stroke at six-month follow up.

Sample size:

Based on determining the main outcome variable, the estimated minimum required sample size is 72 patients (36 patient in each group) .

The sample was calculated using G*power software 3.1.9.2., based on the following assumptions: Main outcome variable is the difference between mean value of MACE rate ( major adverse cardiovascular event) in addict patients undergoing PCI ( percutaneous coronary intervention ) .

Based on clinical experience we expected to find medium effect size difference between 2 groups(addict and non addict patients).

Main statistical test is independant t-test to detect the difference between the 2 groups Alpha = 0.05 Power = 0.90 Effect size = 0.7

Statistical analysis:

Data entry and analysis will be carried out using SPSS version 20. Descriptive statistics will be done, and then analytical statistics will be chosen according to the type of variables. Values will be considered significant when P values less than 0.05

ELIGIBILITY:
Inclusion Criteria:

* All patients of all categories of ages who will be presented with acute coronary syndrome in Assuit University Hospital .

Exclusion Criteria:

* Pateints presented with cardiogenic shock

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all patients presented with acute coronary syndrome in Assuit University Hospital .
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Left ventricular systolic dysfunction in patients presenting with acute coronary syndrome | baseline
  Left ventricular systolic dysfunction is a common and serious complication of acute coronary syndrome that leads to increased risks of sudden death and of heart failure .
  in this study it will be measured using speckle tracking echocardiography.
Thrombolysis in Myocardial Infarction (TIMI) in patients undergoing PCI | baseline
  The TIMI Coronary Grade Flow is an effective and well-studied grading system of coronary reperfusion on an angiogram.
  Grade 0 means complete occlusion of the infarct-related artery Grade 1 means some penetration of contrast material beyond the point of obstruction but without perfusion of the distal coronary bed Grade 2 means perfusion of the entire infarct vessel into the distal bed but with delayed flow compared with a normal artery Grade 3 means full perfusion of the infarct vessel with normal flow

CONTACTS AND LOCATIONS:
Overall Officials: Hossam El Araby, professor, Principal Investigator; Salma Taha, doctor, Principal Investigator